CLINICAL TRIAL: NCT02808416
Title: Personalized Cellular Vaccine Therapy in Treating Patients With Brain Metastases From Solid Tumors
Brief Title: Personalized Cellular Vaccine for Brain Metastases (PERCELLVAC3)
Acronym: PerCellVac3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong 999 Brain Hospital (Other)
Collaborators: Beijing Tricision Biotherapeutics Inc (Industry); Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry); Jinan University Guangzhou (Other)
Responsible Party: Principal Investigator, Jian Zhang, Vice President of the hospital and Chief Physician, Guangdong 999 Brain Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ag-mRNA-Cell-BM-999Brain
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Brain Cancer; Neoplasm Metastases
Keywords: Solid tumors; Brain metastases; DC vaccine; Personalized vaccine; Tumor antigens
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Personalized cellular vaccine (Experimental): Patients will undergo tumor resection or biopsy, and receive biweekly cellular vaccines consisting of mRNA-pulsed autologous DCs.
  Interventions: Biological: Personalized cellular vaccine

INTERVENTIONS:
Biological: Personalized cellular vaccine — Cancer patients with brain metastases will undergo tumor resection or biopsy, and receive tumor antigen mRNA pulsed cellular vaccines.
  Other Names:
  • Tumor antigen pulsed DC and PBMC, autologous tumor vaccine

SUMMARY:
Cancer patients with brain metastases (BM) have poor prognosis. Current treatments produce limited efficacy. Recent advance in cancer immunotherapy has provided important new means to treat cancer patients at advanced stages. This study is designed to perform a clinical trial to treat advanced caner patients with brain metastases with personalized dendritic cell-based cellular vaccines. The patients will receive vaccines consisting of mRNA tumor antigen pulsed DCs. Immune response to the immunized tumor antigens will be monitored. Safety and efficacy will be observed in this study.

DETAILED DESCRIPTION:
This is an open label, single-arm, single-institution, Phase I study designed to investigate the safety and efficacy of personalized cellular tumor vaccines for cancer patients with brain metastases (BM). BM patients will undergo tumor resection or biopsy and the tumor tissues will be analyzed for the expression of tumor antigens and immune-related genes. The patients will be immunized with DCs pulsed with mRNA encoded tumor antigens. Patients will be immunized with DC vaccines on a biweekly basis. Safety and efficacy will be monitored. The objective of this study is to assess the safety of the personalized cellular vaccines and to deterimine the antitumor specific T cell responses. The efficacy of the vaccines will be determined using RANO-BM criteria, progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor with brain metastases.
* Patients at the age of 18-65.
* Patients undergo tumor resection or biopsy.
* Patients with Karnofsky scores > or =70
* Patients with normal range of hematologic and metabolic test results.
* Patients must have no corticosteroids treatment at least one week before vaccination.
* Patients capable of understanding the study and signed informed consent.

Exclusion Criteria:

* Infectious diseases HIV, HBV, HCV.
* Documented immunodeficiency.
* Documented autoimmune disease.
* Breast feeding females.
* Pregnant women.
* Any serious or uncontrolled medical or psychiatric conditions, for example, severe pulmonary, cardiac or other systemic disease.
* Patient inability to participate as determined by PI discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events and severe adverse events (safety and tolerability) | 3 years since the beginning of the first vaccine
  Incidence of adverse events and severe adverse events to measure safety and tolerability of mRNA-TAA pulsed autologous DC vaccines.

SECONDARY OUTCOMES:
Antitumor specific T cell response | 4 weeks after the last vaccine
  The frequency of the peripheral CD8+ and CD4+ T cell response to the vaccine will be measured.
Progression-free survival | 24 months since the beginning of the first vaccine
  Progression-free survival will be monitored for 2 year
Overall survival | 3 years since the beginning of the first vaccine
  Overall survival will be monitored for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, M.D., Principal Investigator — Guangdong 999 Brain Hospital
Locations (1):
- Guangdong 999 Brain Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wang QT, Nie Y, Sun SN, Lin T, Han RJ, Jiang J, Li Z, Li JQ, Xiao YP, Fan YY, Yuan XH, Zhang H, Zhao BB, Zeng M, Li SY, Liao HX, Zhang J, He YW. Tumor-associated antigen-based personalized dendritic cell vaccine in solid tumor patients. Cancer Immunol Immunother. 2020 Jul;69(7):1375-1387. doi: 10.1007/s00262-020-02496-w. Epub 2020 Feb 20. PMID 32078016
- See also: Clinical trial results — https://pubmed.ncbi.nlm.nih.gov/32078016/